CLINICAL TRIAL: NCT07078565
Title: Comparative Effects of Tai Chi Versus Modified-Otago Exercises On Pain, Balance And Motor Function In Patients With Diabetic Peripheral Neuropathy
Brief Title: Tai Chi vs. Modified-Otago Exercises for Pain, Balance, and Motor Function in Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0295
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy (DPN); Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetic Peripheral Neuropathy; Tai Chi; Modified-Otago Exercises; Balance Training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi (Experimental): Participants in this group will receive Tai Chi-based therapeutic exercise sessions, including joint mobility, balance, flexibility, and strength training movements (e.g., Qigong and bow stance).
  Interventions: Other: Tai Chi
- Modified-Otago Exercises (Experimental): Participants in this group will receive the Modified-Otago Exercise Program focused on strength and balance training through functional exercises like stair walking, knee bends, and toe raises.
  Interventions: Other: Modified-Otago Exercises

INTERVENTIONS:
Other: Modified-Otago Exercises — Intervention is administered 3 times per week for 4 weeks, with the same baseline therapy as the Tai Chi group.
  Arms: Modified-Otago Exercises
Other: Tai Chi — Intervention is administered 3 times per week for 4 weeks, along with baseline therapy (TENS + heating pad).
  Arms: Tai Chi

SUMMARY:
his randomized clinical trial evaluates the comparative effectiveness of Tai Chi and Modified-Otago exercise programs on pain reduction, balance improvement, and motor function in patients diagnosed with diabetic peripheral neuropathy (DPN). DPN is a common complication of Type 2 Diabetes Mellitus that significantly impairs quality of life through chronic pain, balance deficits, and decreased functional mobility. While pharmacological treatments are commonly used, they often result in adverse side effects, creating a growing need for non-pharmacological interventions like therapeutic exercises.

Tai Chi, a traditional Chinese exercise combining slow movements and mental focus, has shown benefits in improving mobility and reducing fall risks in chronic disease populations. The Modified-Otago program, originally developed to prevent falls in the elderly, emphasizes strength and balance training through structured exercise routines.

A total of 36 participants (aged 40-80 years) with at least a 5-year history of Type 2 diabetes and a minimum pain score of ≥3 on the Numeric Pain Rating Scale (NPRS) will be recruited. Participants will be randomly allocated to either the Tai Chi group or the Modified-Otago group. Both groups will receive 24 sessions over an 8-week period (3 sessions per week), along with baseline interventions such as heating pad application, TENS, and warm-up/cool-down routines.

Primary outcome measures include NPRS for pain, the Berg Balance Scale (BBS) for balance, and the Dynamic Gait Index (DGI) for motor function. Assessments will be conducted at baseline, post-intervention, and two weeks post-treatment. Data will be analyzed using SPSS version 26 to determine within-group and between-group differences.

This study aims to inform clinicians about effective exercise strategies for improving physical function in patients with DPN and potentially establish evidence-based rehabilitation protocols.

DETAILED DESCRIPTION:
Diabetic Peripheral Neuropathy (DPN) is a chronic complication of diabetes characterized by pain, numbness, and impaired balance. It frequently leads to limitations in mobility and increased fall risk, significantly affecting patients' independence and quality of life. Standard treatments often include pharmacological agents, but their long-term use is associated with adverse effects. As a result, non-drug interventions like exercise are increasingly being promoted as safer and equally effective alternatives.

Tai Chi and Modified-Otago exercise programs have individually shown promise in populations with mobility impairments. Tai Chi integrates slow, controlled movements with breathing and mindfulness, making it suitable for elderly individuals or those with chronic conditions. The Modified-Otago program was specifically designed to prevent falls through strength and balance training. While both interventions are beneficial independently, no study has yet compared their relative efficacy in managing symptoms of DPN.

ELIGIBILITY:
Inclusion Criteria:

* Both genders are aged 40-80 years
* Patient having Types ii diabetes with Minimum of 5 years since diabetes diagnosis
* Patients experiencing chronic pain for at least 6 months and level ≥ 3 on NPRS.
* Patient having ≥ 6 score on Toronto Clinical Neuropathy Scoring System for diabetic neuropathy

Exclusion Criteria:

* Non-ambulatory patients
* Patients with ulceration/infection of feet, medical/surgical conditions
* Patients suffering from stroke, parkinson's disease, or multiple sclerosis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), which rates pain on a scale from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Balance | 4 weeks
  Balance will be assessed using the Berg Balance Scale (BBS), a 14-item scale that evaluates static and dynamic balance in older adults.
Gait Performance | 4 weeks
  Motor function and dynamic walking ability will be measured using the Dynamic Gait Index (DGI), which assesses an individual's ability to modify gait in response to changing task demands.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab Training and Research Center,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to institutional policies, ethical considerations, and privacy concerns. All data will be kept confidential and used solely for the purposes of this stud